CLINICAL TRIAL: NCT06204666
Title: Influence of 2-Weeks Hemp Fiber Ingestion on Gut Permeability and Metabolite Shifts After Vigorous Exercise
Brief Title: Hemp Fiber Ingestion and Gut Permeability After Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HS-24-86
Record Dates: First submitted 2023-12-19; First posted 2024-01-12 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Gastrointestinal Dysfunction; Metabolic Disturbance
Keywords: hemp fiber; exercise; gut permeability; metabolomics
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized treatment, double blinded procedures, crossover
Who Masked: Participant, Investigator
Masking Description: Investigators and study participants will be blind to treatment allocation, with the hemp fiber-based supplement bars and placebo supplement bar of the same texture, taste, and look.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Dose Hemp Fiber Bar (Experimental): 20% hemp hull powder
  Interventions: Dietary Supplement: High Dose Hemp Fiber Bar
- Low Dose Hemp Fiber Bar (Experimental): 5% hemp hull powder
  Interventions: Dietary Supplement: Low Dose Hemp Fiber Bar
- Placebo (Placebo Comparator): 0% hemp hull powder
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: High Dose Hemp Fiber Bar — High dose hemp fiber bar with other ingredients
  Arms: High Dose Hemp Fiber Bar
Dietary Supplement: Low Dose Hemp Fiber Bar — Low dose hemp fiber bar with other ingredients
  Arms: Low Dose Hemp Fiber Bar
Dietary Supplement: Placebo — Placebo bar with other ingredients
  Arms: Placebo

SUMMARY:
Two bioactive compounds, N-trans-caffeoyl tyramine (NCT) and N-trans-feruloyl tyramine (NFT), have been investigated for potential gut health benefits. The shells of hemp seeds are a rich source of NCT and NFT. The hypothesis for this project is that ingestion of a hemp fiber bar containing NCT and NFT will mitigate exercise-induced increases in gut permeability. This study will examine the efficacy of 2-weeks ingestion of a hemp fiber bar (high and low doses) in moderating exercise-induced gut permeability using a randomized crossover trial.

Objective #1: To conduct a randomized crossover trial using placebo-controlled, double-blind procedures with 20 cyclists who will in random order ingest a hemp fiber bar supplement (high and low doses) or placebo each day for two weeks prior to an exercise challenge (2.25 hours of intensive cycling).

Objective #2: To determine if hemp fiber bar supplementation attenuates exercise-induced gut permeability using several outcome measures including plasma lactulose to 13C mannitol (L:M) ratio and plasma intestinal fatty acid binding protein (I-FABP) as markers of gastrointestinal permeability and mucosal damage, respectively. Shifts in thousands of metabolites will be measured via untargeted metabolomics to provide additional gut permeability biomarkers and help reveal underlying mechanisms.

DETAILED DESCRIPTION:
This study will employ a randomized crossover design. Study participants will be block randomized to three trials (high and low dose hemp fibers bars or placebo) using double-blinded, placebo-controlled procedures. The supplement bars will be coded by the sponsor, with the double-blind code held until after all study samples have been analyzed. Subjects will come to the lab for orientation/baseline testing, pre-and post-supplementation blood sample collections (2 weeks supplementation with high and low dose hemp fiber bar supplements or placebo), and three 2.25 h cycling sessions (thus 9 total lab visits).

A. Orientation (Visit #1). Subjects will report to the lab in an overnight fasted state. Subjects will voluntarily sign IRB-approved consent forms and complete questionnaires (delayed onset of muscle soreness or DOMS, Profile of Mood States or POMS). Demographic, health, and training histories will be acquired with questionnaires. A blood sample will be collected. Subjects will ingest a standardized sugar solution containing lactulose 5 g, 13C mannitol 100 mg, mannitol 1.9 g, and rhamnose 1 g in a total of 450 ml water (SS, calculated osmolality 69 mosmol/kg). An increase in the post-exercise lactulose/13C mannitol ratio (L/M) will be used as an indicator of increased gut permeability. All urine excreted from 0-5 h post SS ingestion will be collected in a urine collection container. Subjects will be urged to drink water after the first hour of the test to ensure adequate urine output. The Boost beverage will be consumed at 7 kcal/kg 1.5 h post SS ingestion (to simulate what occurs post-exercise). The urine collection container will be placed in the refrigerator until they are returned to the lab the next day. The total urine volume will be measured with four 50 ml aliquots frozen in a minus 80°C freezer until analysis.

B. Baseline Testing/Pre-Supplementation (Visit #2). Subject will return urine collection container to the HPL the day after Visit #1. Body composition will be measured with the seca BIA and Bod Pod body composition analyzer (Life Measurement, Concord, CA). Study participants will be tested for maximal aerobic capacity (VO2max) during a graded, cycling test with continuous metabolic monitoring with the Cosmed CPET metabolic device (Cosmed, Rome, Italy). A 2-week supply of high dose or low dose hemp fiber bars or placebo bars will be given to the participants. Subjects will consume 2 bars per day, one with the first meal in the morning and the second bar with the last meal of the day.

C. 2.25 h Cycling Session (Lab Visit #3): During the 3-day period prior to the 2.25-h cycling session, subjects will taper exercise training and ingest a moderate-carbohydrate diet using a food list restricting high fat foods, visible fats, and caffeine. Subjects will record all food and beverage intake in a 3-day food record with macro- and micro-nutrient intake calculated using the ESHA Food Processor nutrient analysis software program. Study participants will report to the Human Performance Lab in an overnight fasted state and provide a blood sample, ingest the supplement (1 hemp fiber bar or placebo bar), and then cycle 2.25 h at high intensity (70% VO2max) while ingesting water alone (3 ml/kg every 15 minutes). Immediately following the cycling bout, subjects will ingest the SS. Blood samples will be collected at 0 h, 1.5 h, and 3.0 h post-exercise. All urine excreted from 0-5 h after SS ingestion will be collected in a urine collection container.

Testing protocol during the lab sessions with the 2.25-h cycling session:

1. 7:00 am: Provide blood sample, DOMS rating (1-10 scale), and POMS. Complete the symptom survey. Turn in the 3-day food record.
2. 7:10 am: Ingest 1 supplement bar with 1 cup water.
3. 7:30 am: Start the 2.25 h cycling session. Subjects will cycle on trainers at 70% VO2max (~race pace) for 2.25 hours. Oxygen consumption, carbon dioxide production, respiratory exchange ratio, and ventilation will be measured using the Cosmed Quark CPET metabolic cart every 30 minutes. Subjects will consume 3 ml/kg water every 15 min. No other beverage or food containing energy or nutrients will be allowed during the 2.25-h exercise sessions.
4. ~10:00 am to 1:00 pm: Ingest the 450 mL SS within the first minute of getting off the bicycle. All urine excreted from 0-5 h after SS ingestion will be collected in a urine collection container. Blood samples will be taken via venipuncture immediately after completing the cycling session, and then 1.5-h and 3.0-h post-exercise. Subjects will be allowed to shower and change clothes. The DOMS and POMS questionnaires will be administered each time blood samples are collected. Subjects will ingest no food or beverage other than water (7 ml/kg during the 1.5 h post-exercise period; this will take into account the 450 ml sugar solution; no water will be ingested during the first hour post-SS intake). After the 1.5 h post-exercise blood draw, subjects will ingest a Boost beverage (7 kcal/kg body weight). Another blood sample will be collected 3-h post-exercise. Afterwards, subjects will be allowed to stay in the lab to complete the 5h urine collection (preferred procedure) or leave the lab and return later in the day to turn in the 5h urine container. Upon request, subjects can also leave the lab, finish the 5h urine collection, put the container in the refrigerator, and then bring the urine container to the lab the next morning.

D. Washout/Crossover/Repeat

Subjects will engage in a 2-week washout period without the supplements, crossover to the next treatment arm, and then repeat all procedures except for the consent process, completion of the medical health questionnaire, body composition testing, and VO2 max testing (Lab visits #4,5,6). Subjects will maintain the study diet and normal exercise training routines during the 2-week washout period.

E. SECOND Washout/Crossover/Repeat

Subjects will engage in a 2-week washout period without the supplements, crossover to the next treatment arm, and then repeat all procedures except for the consent process, completion of the medical health questionnaire, body composition testing, and VO2 max testing (Lab visits #7,8,9).

ELIGIBILITY:
Inclusion Criteria:

* Male or female cyclists, ages 18-65 years, and capable of cycling 2.25 h in the laboratory at 60% watts maximum (close to long-distance race pace).
* Non-smoker, and generally healthy and without gastrointestinal diseases (irritable bowel syndrome, chronic nausea, vomiting, and diarrhea, Crohn's disease, Celiac disease, diverticulosis) or chronic diseases including cardiovascular disease (e.g., heart disease, stroke), cancer, type 1 and 2 diabetes, rheumatoid arthritis. Categorized as "low risk" using the American College of Sports Medicine screening questionnaire.
* Agree to train normally, maintain weight, and avoid the regular use of large-dose vitamin and mineral supplements, herbs, and medications that influence inflammation (especially non-steroidal antiinflammatory drugs or NSAIDs) for the duration of the 10-week study and at least a 2-week period prior to the study.
* Agree to taper your exercise routine prior to each of the 3 lab cycling sessions (as if preparing for a race event).
* Agree to restrict (i.e., avoid high amounts of) black pepper, red pepper, garlic, curry, and other strong spices during the 3-day period prior to each lab visit.

Exclusion Criteria:

* Inability to comply with study requirements.
* Females trying to become pregnant, or currently pregnant or breastfeeding.
* Nonpregnant adults who weigh less than 110 pounds.
* Any other concurrent condition which, in the opinion of the principal investigator (PI), would preclude participation in this study or interfere with compliance.
* Current diagnosis of gastrointestinal disease, cardiovascular disease, diabetes, or cancer (except for non-melanoma skin cancer).
* Sensitivity to hemp fiber.
* History of intolerance to cow's milk and lactose.
* History of adverse symptoms to low amounts of lactulose, mannitol, and rhamnose sugars (low calorie and poorly absorbed sugars).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-12-09 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Gut permeability | Change from pre-supplementation levels to 5 hours post-exercise
  Urine concentrations of post-exercise lactulose/13C mannitol ratio (L/M)

SECONDARY OUTCOMES:
Changes in plasma hemp fiber-related metabolites including acetic acid, propionic acid, and butyric acid from targeted metabolomics using LC-MS/MS analysis (relative intensities) | Change from pre-study to post-2 weeks supplementation, and immediately post-exercise, and 1.5 hours-, 3 hours-, and 24 hours-post-exercise
  Targeted metabolomics to assess plasma metabolites (short chain fatty acids) from LC-MS/MS analysis (relative intensities)

CONTACTS AND LOCATIONS:
Overall Officials: David C Nieman, DrPH, Principal Investigator — Appalachian State University
Locations (1):
- Appalachian State University Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share data upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: January 2024, indefinitely
Access Criteria: Will share information upon reasonable request.